CLINICAL TRIAL: NCT02501551
Title: A Phase II Study to Evaluate the Efficacy of Regorafenib in C-kit Mutated Metastatic Malignant Melanoma Failed First-Line Dacarbazine, Temozolomide or Immune Therapy
Brief Title: Regorafenib, C-kit Mutated Malignant Melanoma, 2nd Line Therapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Principal Investigator, Sang Joon Shin, Associate Professor, Yonsei University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4-2014-0573
Record Dates: First submitted 2015-03-05; First posted 2015-07-17 (Estimated); Last update posted 2021-04-05 (Actual); Status verified 2021-04

CONDITIONS: Melanoma
Keywords: Malignant melanoma; C-KIT mutation
MeSH Terms: conditions — Melanoma | interventions — regorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Regorafenib (Experimental): 160mg regorafenib once daily with a low fat breakfast for the first 21 days of each 28-day cycle
  Interventions: Drug: regorafenib

INTERVENTIONS:
Drug: regorafenib — 160mg regorafenib once daily with a low fat breakfast for the first 21 days of each 28-day cycle

SUMMARY:
This is a phase II trial of regorafenib in patients with metastatic melanoma harboring c-Kit mutations and/or amplifications of c-Kit gene copy number. The primary end point is disease control rate (DCR), and the secondary end points are safety, response rate (RR), progression free survival (PFS), and overall survival (OS).

DETAILED DESCRIPTION:
The incidence of melanoma is rising globally and mortality is increasing faster than most other cancers. Recent advances in the molecular biology of melanoma have uncovered several potential therapeutic targets in melanoma. It has been observed that 81% of melanomas arising from non-chronic sun-damaged skin have an oncogenic BRAF or NRAS mutation, whereas such mutations are far less frequent in chronic sun-damaged skin melanomas, acral melanomas, or mucosal melanomas. In contrast, c-Kit mutations are more common in mucosal and acral melanomas, which can also be accompanied by an increase in c-Kit copy numbers.

Asian populations, the most common melanoma subtypes are acral and mucosal melanoma, which comprise greater than 70% of all melanomas, a rate that is much higher than that seen in white populations (6% to 7%). KIT mutations or amplification are reported about 20% in acral or mucosal melanomas (JAMA. 2011;305(22):2327-2334). Therefore, c-Kit mutations are likely the most common kind of genetic mutations in Asians, and the investigation of c-Kit inhibitors is a high priority in this population.

Imatinib mesylate (Gleevec, formerly STI571; Novartis Pharmaceuticals, Basel, Switzerland), is a selective inhibitor, targeting Abl as well as c-Kit and the platelet-derived growth factor receptor. Imatinib demonstrated significant activity in patients with metastatic melanoma harboring genetic c-Kit aberrations, with an overall response rate of 29% (J Clin Oncol 2011;29:2904-9) Regorafenib (BAY 73-4506) is a novel, orally active, diphenylurea multikinase inhibitor of VEGFR1-3, c-KIT, TIE-2, PDGFR-β, FGFR-1, RET, RAF-1, BRAF and p38 MAP kinase. Regorafenib provide a significant improved PFS and OS in patients with GIST and colorectal cancer, respectively (Lancet 2013; 381: 295-302, Lancet 2013; 381: 303-12). Especially, inhibitory activity of regorafenib is most effective in c-kit mutated tumors. Therefore, regorafenib has a chance to significant activity in melanoma with c-kit mutations. However, no clinical trials have been published for regorafenib in the patients with melanoma who harbor c-Kit mutations.

NCCN recommend ipilimumab, high-dose interleukin-2, and vemurafenib or dabrafenib for BRAF mutated tumor as a preferred regimen, and imatinib for c-kit mutated tumors, dacarbazine, temozolomide, and paclitaxel as other active regimens. In Korea, ipilimumab is not available yet and imatinib for c-kit mutated tumors is not used legally. Thus, regorafenib could be used for c-kit mutated tumor in clinical trial setting.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically proven melanoma with stage IV or unresectable stage III disease
2. c-kit mutations
3. performance status of 0, 1, and 2
4. Have progressed after 1 previous systemic treatment containing dacarbazine, temozolomide, or immunotherapy for metastatic melanoma
5. Patients with central nervous system metastasis must have stable neurologic function without evidence of central nervous system progression within 8 weeks
6. Measurable disease or non-measurable but evaluable disease, according to the Response Evaluation Criteria in Solid Tumors v1.1

Exclusion Criteria:

1. Major surgery or radiation therapy within 4 weeks of starting the study treatment
2. History of or known carcinomatous meningitis, or evidence of symptomatic leptomeningeal disease
3. Have received greater than or equal to 2 previous chemotherapy-containing systemic treatment regimens
4. Patients with BRAF or NRAS mutation
5. Prior therapy with a c-kit inhibitor
6. Significant history of cardiac disease, myocardial infarction, or current cardiac ventricular arrhythmias requiring medication
7. Major surgery within 4 weeks before start of study treatment
8. Active gastrointestinal bleeding
9. Patients treated with co-administration of a strong CYP3A4 inducers
10. Adequate Hematologic, Biochemical, and Organ Function

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2015-02; Primary Completion 2022-05 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
disease control rate as measured by RECIST 1.1 | at 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Yonsei University Health System, Seoul, South Korea